CLINICAL TRIAL: NCT05948241
Title: Online Psychological Support Group for Patients With Heart Failure and Depression in Promoting Self-care: a Randomized Clinical Trial
Brief Title: Online Psychological Support Group for Patients With Heart Failure and Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UP 5977/21
Record Dates: First submitted 2023-06-21; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-06

CONDITIONS: Heart Failure; Depression
MeSH Terms: conditions — Heart Failure; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment (Active Comparator): The control group will undergo 1 consultation with the multidisciplinary team, offered as standard treatment at the Heart Failure outpatient clinic of the Institute of Cardiology, with the areas: medicine, nutritionist and psychology. Monitoring with a multidisciplinary team is the gold standard for monitoring patients with HF and its multiple comorbidities. These patients are followed up on average every 3 months in this outpatient clinic.
  Interventions: Other: Standard multidisciplinary care
- Online psychological support group (Experimental): The intervention group, in addition to standard treatment, will have 1 weekly session in an online psychological support group of 45 minutes each, totaling 12 sessions in three months. The intervention will be carried out by research psychologists specializing in cardiology, with online consultations via whatsapp
  Interventions: Other: Online psychological support group

INTERVENTIONS:
Other: Online psychological support group — 1. st Session: Presentation of the participants and the objectives of the group, which are the management of depression and the promotion of self-care. Discussion on heart failure and its clinical management. Arrangements will be made with these patients about confidentiality between the participants, as it is a group intervention where each participant can expose their personal issues.
  2. nd Session: Discussion on depression and its clinical management. From the 3rd to the 11th Session: They will aim to offer support for the emotional demands of the participants, related to the daily and future challenges inherent in the care provided with HF, seeking to promote self-care. As it is a homogeneous group, it is expected to enable enriching exchanges within the group about changes in habits or adaptations to HF, since psychological support groups have this function.
  12th Session: Closing and evaluation of participants. Scheduling for reassessment of instruments
  Arms: Online psychological support group
Other: Standard multidisciplinary care — The control group will undergo 1 consultation with the multidisciplinary team, offered as standard treatment at the Heart Failure outpatient clinic of the Institute of Cardiology, with the areas: medicine, nutritionist and psychology. Monitoring with a multidisciplinary team is the gold standard for monitoring patients with HF and its multiple comorbidities. These patients are followed up on average every 3 months in this outpatient clinic.
  Arms: Standard treatment

SUMMARY:
Heart failure is a chronic disease, being the second cause of death in Brazil. Currently, it is estimated that 6.4 million Brazilians suffer from this disease. The higher number of rehospitalization, lower survival of these individuals. There are recommendations from Societies of Cardiology for the inclusion of effective self-care for patients with chronic HF, intend greater control of symptoms, greater adherence to treatment and, consequently, decrease of rehospitalization. One of the pillars of self-care's education for chronic patients recommended by the Health Ministry is the management of the patient's emotional aspects. These have been undertreated in most studies. The prevalence of depression among patients with HF is high and ranges from 41% to 72%, and the assessment with the BDI-II, which is the gold standard used, is 67%. Patients with HF and depression have greater difficulty in adhering to treatment and poor maintenance of self-care. Also, they present 4 times more risk of rehospitalization/mortality. Faced with this problem, this project was designed, proposing an online psychological support group for patients with heart failure and depression, primarily aimed at improving self-care, adherence and secondarily at reducing the rates of depression and readmission.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with heart failure
* Age between 18 and 79 years B)
* After hospital discharge
* Depression (BDI-II score above 14 points)
* Acceptance of the Term of Consent;

Exclusion Criteria:

* Patients with dementia
* Communication barriers
* Octogenarians
* People unable to access the internet for the intervention
* Who declined to participate;

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 132 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2023-12-05 (Estimated)

PRIMARY OUTCOMES:
Changes in European Heart Failure Self-Care Behavior Scale's Scores | From baseline to 4 months
  Changes in Self-care scale scores

SECONDARY OUTCOMES:
Changes in Beck Depression Inventory Scores (BDI-II) | From baseline to 4 months
  Changes in depression scores
Changes in Morisky and Green points | From baseline to 4 moths
  Changes in adherence points
The average hospitalization's days in 1 year follow up | From baseline to 1 year follow up
  The average hospitalization days in 1 year follow up for all causes heart failure related

CONTACTS AND LOCATIONS:
Overall Officials: MARCIA M SCHMIDT, Principal Investigator — IC-FUC
Locations (1):
- Marcia Moura Schmidt, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No